CLINICAL TRIAL: NCT00018005
Title: Heart Failure Adherence and Retention Trial (HART)
Brief Title: A Self-Management Intervention for Mild to Moderate Heart Failure
Acronym: HART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lynda Powell, PhD, MEd (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Lynda Powell, PhD, MEd, Chair, Department Preventive Medicine, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 137; R01HL065547 (NIH)
Record Dates: First submitted 2001-06-26; First posted 2001-06-26 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure, Congestive
Keywords: Heart Failure; Self-Management; Behavioral Clinical Trial
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure | interventions — Self-Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Self-Management — 18 in-person group sessions providing self-management training.
Other: attention control — 18 educational mailings follow by a a telephone call.

SUMMARY:
This study will test whether a self-management (SM) intervention, compared to usual care, will reduce the risk for adverse clinical outcome in patients with mild to moderate heart failure.

DETAILED DESCRIPTION:
BACKGROUND:

Heart failure is a major disabling disease for American adults, affecting an estimated 4.9 million individuals. Heart failure is associated with enormous health care expenditures. This is because it is a progressive chronic condition that is characterized by disabling symptoms that limit independence and result in multiple hospitalizations and referrals to long-term care. The emergence of heart failure as a major public health problem is related to the unintended result of both an aging population and the success in reducing mortality from cardiovascular disease. Non-adherence to medications is a key problem in the treatment of heart failure, with adherence rates ranging from 20% to 90%. There is a clear need, therefore, to develop interventions that improve adherence in patients with heart failure.

DESIGN NARRATIVE:

This is a single-site, partially blinded, randomized clinical trial of 900 patients with systolic or diastolic dysfunction, and New York Heart Association (NYHA) functional class II or III. Patients will be recruited over a period of 2 years from seven hospitals. Patients will be randomly assigned to either a SM intervention or attention control. The SM group will meet 18 times for 2 hours over 1 year. These group sessions will teach patients how to use five basic self-management skills (self-monitoring, environmental restructuring, social support, cognitive restructuring, and the relaxation response) to help build self-efficacy and maintain it after the treatment has been discontinued. The attention control arm will consist of an educational intervention which includes 18 mailings of the American Heart Association Tip Sheets over the course of the first year, plus a telephone follow-up with the patient after each mailing to check receipt and comprehension of the Tip Sheet, and to address any questions about the Tip Sheet. Treatment effects will be evaluated using the primary outcome of hospitalization for heart failure or death, and the secondary outcomes of progression of heart failure, quality of life, and health care costs. Potential mediators of effectiveness will include improved adherence and improved psychosocial function.

ELIGIBILITY:
Inclusion Criteria:

* NYHA classification of II or III
* LVEF of 40% or less

Exclusion Criteria:

* Uncertain 12-month prognosis
* Potential cardiac transplant within 1 year of study entry
* Severe aortic stenosis
* Uncontrolled ventricular tachycardia
* Non-cardiac causes of heart failure symptoms (i.e., peripheral vascular disease, chronic obstructive pulmonary disease, and arthritis)
* Major psychiatric co-morbidity
* Unstable angina, myocardial infarction, coronary artery bypass graft, or percutaneous transluminal coronary angioplasty within 1 month prior to study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2001-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time until all-cause death or heart-failure hospitalization | Measured over the two years of study follow-up.
  This is a composite outcome, measuring time from randomization to occurrence of death due to any cause or a hospitalization that is adjudicated to be due to heart-failure, among participants who experience either (or both) of these events. Only the first occurrence of either of these events is considered.

SECONDARY OUTCOMES:
Progression of heart failure | Measured over the two years of study follow-up
  Measured using change in NYHA Class and Six-Minute Walk distance, from baseline.
Quality of life | Measured over the two years of study follow-up
  Measured using self-report heart-failure-specific quality of life scales.
Health care costs | Measured over the two years of study follow-up
Time until all-cause death or all-cause hospitalization | Measured over the two years of study follow-up
  This is a composite outcome, measuring time from randomization to occurrence of death due to any cause or hospitalization for any reason, among participants who experience either (or both) of these events. Only the first occurrence of either of these events is considered.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda H. Powell, Study Chair — Rush-Presbyterian-St. Lukes Medical Center
Locations (1):
- Rush-Presbyterian-St. Lukes Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Doukky R, Mangla A, Ibrahim Z, Poulin MF, Avery E, Collado FM, Kaplan J, Richardson D, Powell LH. Impact of Physical Inactivity on Mortality in Patients With Heart Failure. Am J Cardiol. 2016 Apr 1;117(7):1135-43. doi: 10.1016/j.amjcard.2015.12.060. Epub 2016 Jan 18. PMID 26853954
- [Derived] Doukky R, Avery E, Mangla A, Collado FM, Ibrahim Z, Poulin MF, Richardson D, Powell LH. Impact of Dietary Sodium Restriction on Heart Failure Outcomes. JACC Heart Fail. 2016 Jan;4(1):24-35. doi: 10.1016/j.jchf.2015.08.007. PMID 26738949
- [Derived] Powell LH, Calvin JE Jr, Richardson D, Janssen I, Mendes de Leon CF, Flynn KJ, Grady KL, Rucker-Whitaker CS, Eaton C, Avery E; HART Investigators. Self-management counseling in patients with heart failure: the heart failure adherence and retention randomized behavioral trial. JAMA. 2010 Sep 22;304(12):1331-8. doi: 10.1001/jama.2010.1362. PMID 20858878
- [Derived] Powell LH, Calvin JE Jr, Mendes de Leon CF, Richardson D, Grady KL, Flynn KJ, Rucker-Whitaker CS, Janssen I, Kravitz G, Eaton C; Heart Failure Adherence and Retention Trial Investigators. The Heart Failure Adherence and Retention Trial (HART): design and rationale. Am Heart J. 2008 Sep;156(3):452-60. doi: 10.1016/j.ahj.2008.05.011. PMID 18760125